CLINICAL TRIAL: NCT00168142
Title: MVCT Imaging Pilot Study Using Helical Tomotherapy
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 21131
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-12

CONDITIONS: Cancer, Carcinoma
Keywords: Helical tomotherapy; Megavoltage imaging
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare the two types of scans, the conventional CT planning scan and the tomotherapy planing scan.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing radiotherapy metallic artifact in radiation field.

Exclusion Criteria:

* Contraindication to radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2003-10; Primary Completion 2008-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rufus Scrimger, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada